CLINICAL TRIAL: NCT01205763
Title: Evaluation of Effects of Clavicular Hook Plate on Subacromial Space
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wei-Pin Ho, Department of Orthopaedics
Other Study IDs: 98086
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: AC Joint Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators intend to demonstrate that the hook plate may have adverse effects on subacromial structures even with a short period of hardware retention. The investigators also sought to determine if musculoskeletal sonography could be used as a tool to demonstrate shoulder pathology such as subacromial impingement or rotator cuff tear in patients receiving hook plate fixation. The clinical results of patients receiving hook plate fixation, specifically bony union, pain relief, shoulder function and range of motion (ROM), were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient received surgical treatment for AC joint dislocation of unstable distal clavicle fracture in our hospital from December 2007 to January 2009.

Exclusion Criteria:

* The patient who was expired or the injured limb has preexisting injury or neurological deficit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient received surgical treatment for AC joint dislocation of unstable distal clavicle fracture
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-12; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Pin Ho, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan